CLINICAL TRIAL: NCT07176819
Title: Effectiveness of Gait Retraining in Female Runners With Patellofemoral Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Gait Retraining in Female Runners With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 277H
Record Dates: First submitted 2025-09-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2023-03

CONDITIONS: Patellofemoral Pain, PFP
Keywords: Patellofemoral pain; gait retraining
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait retraining group (Experimental): Participants received a 6-week gait retraining program plus patient education. The gait retraining program primarily consisted of increasing the step rate by 10%, monitored via a smartwatch.
  Interventions: Behavioral: Gait retraining; Behavioral: Education
- Control group (Active Comparator): Participants received a 6-week patient education program, which included PFP education, load management strategies, symptom-based training modifications, and strengthening exercises.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Gait retraining — The intervention is a wearable device-assisted gait retraining program designed specifically for female runners with patellofemoral pain (PFP). Unlike conventional physiotherapy or exercise-based interventions, this program integrates real-time biofeedback through a commercially available smartwatch and its mobile application. Participants are instructed to increase their step rate by 10% above their preferred cadence. The smartwatch provides auditory metronome cues and real-time cadence feedback to ensure accurate step-rate modification.
  Arms: Gait retraining group
Behavioral: Education — PFP education, load management strategies, symptom-based training modifications, and strengthening exercises.

SUMMARY:
Patellofemoral pain (PFP) is the most common running-related overuse injury, with prevalence up to 17% among runners. Increased patellofemoral joint stress (PFJS) is a major biomechanical contributor to PFP. Traditional strengthening exercises improve function but do not alter running biomechanics. Gait retraining, particularly cadence modification, has been proposed as a promising approach to reduce PFJS and alleviate symptoms. However, evidence from randomized controlled trials remains limited. This study investigates whether wearable device-assisted gait retraining reduces pain, improves function, and modifies running biomechanics in female runners with PFP compared to education alone.

ELIGIBILITY:
Inclusion Criteria:

* Female, Age 18-45 years
* Unilateral/bilateral anterior knee pain > 4 weeks
* VAS pain ≥ 3/10 during running and ≥ 2 of the following: jumping, squatting, kneeling, stairs, prolonged sitting, or resisted knee extension
* Running ≥ 15 km per week
* Natural rearfoot striker

Exclusion Criteria:

* Acute trauma, history of patellar dislocation, meniscal/chondral lesions
* Prior knee surgery or injection in past 12 months
* Rheumatologic, neurologic, or degenerative disease
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain | Baseline, Week 6, Week 18
  The Visual Analogue Scale (VAS) is a validated, widely used instrument for assessing subjective pain intensity. It consists of a 10-centimeter horizontal line, with one end (0) representing "no pain" and the other end (10) representing "worst imaginable pain."

SECONDARY OUTCOMES:
Anterior Knee Pain Scale | Baseline, Week 6, Week 18
  The Anterior Knee Pain Scale (AKPS), also referred to as the Kujala Score, is a patient-reported outcome measure designed to evaluate symptoms and functional limitations associated with anterior knee pain and patellofemoral disorders. It consists of 13 items covering domains such as pain during various activities (e.g., walking, running, jumping, climbing stairs, squatting), functional limitations, abnormal gait, muscle atrophy, and difficulty with prolonged sitting. Each item is scored on an ordinal scale, and the total score ranges from 0 to 100, with higher scores indicating better knee function and fewer symptoms.
Peak Knee Flexion Angle During Running | Baseline, Week 6
  Peak knee flexion angle will be assessed during running trials using a 3-dimensional motion capture system. Reflective markers will be placed according to a standard lower-limb biomechanical model. The angle is defined as the maximum knee flexion angle observed during stance phase of running.
Ground Reaction Force During Running | Baseline, Week 6
  Ground reaction force (GRF) will be measured during overground running using embedded force plates synchronized with motion capture. The variable of interest is the peak force normalized to body weight.
Running Cadence | Baseline, Week 6
  Running cadence will be assessed as the number of steps taken per minute during running. Measurement will be conducted using a wearable device running sessions
Weekly running distance | Baseline, Week 6
  Weekly running distance will be recorded as the total distance covered in running sessions over a 7-day period. Data will be collected from participants' GPS-based tracking devices.

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Nan Wang, Principal Investigator — Beijing Sport University
Locations (1):
- Beijing Sport University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
- What IPD will be shared: De-identified individual participant data that underlie the results reported in the publication, including baseline characteristics, outcome measures (pain scores, functional scores, running mechanics), and adverse events.
  - When will IPD be available: Beginning 6 months after publication of the main trial results, for up to 5 years.
  - With whom: Researchers who provide a methodologically sound proposal to achieve aims consistent with the original study.
  - For what types of analyses: For individual participant data meta-analyses and reproducibility purposes.
  - How to access data: Proposals should be directed to the corresponding author (wanghaonan@bsu.edu.cn). Data access will be provided via secure data transfer after approval of a data-sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the main trial results, for up to 5 years.
Access Criteria: - With whom: Researchers who provide a methodologically sound proposal to achieve aims consistent with the original study.
  - For what types of analyses: For individual participant data meta-analyses and reproducibility purposes.
  - How to access data: Proposals should be directed to the corresponding author (wanghaonan@bsu.edu.cn). Data access will be provided via secure data transfer after approval of a data-sharing agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT07176819/Prot_SAP_000.pdf